CLINICAL TRIAL: NCT04981327
Title: The API-CALF Study: Apixaban to Treat Calf Vein Thrombosis
Acronym: API-CALF
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Marc Righini, Full professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APICALF
Record Dates: First submitted 2021-07-07; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Deep Vein Thrombosis
Keywords: Isolated distal deep vein thrombosis; Anticoagulation; Direct oral anticoagulants
MeSH Terms: conditions — Venous Thrombosis | interventions — apixaban; Tablets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Strategies to protect against bias include randomization with allocation concealment, enrolling consecutive patients. Patients will be advised to not disclose to study personnel during follow-up to which arm they were randomized to. Adjudicators will be blinded from treatment allocation group, and we will use standardized, validated measures to diagnose DVT, PE, PTS, and bleeding. We plan to allow phone follow-up to limit the risk of lost to follow-up and the impact on patients' in person consultation of a COVID wave during the course of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): After a conventional course of 7 days of Apixaban 10mg BID, Apixaban 2.5mg BID during 3 months.
  Interventions: Drug: Apixaban 2.5 MG Oral Tablet [ELIQUIS]
- Standard (Active Comparator): After a conventional course of 7 days of Apixaban 10 mg BID, Apixaban 5 mg BID during 3 months.
  Interventions: Drug: Apixaban 2.5 MG Oral Tablet [ELIQUIS]

INTERVENTIONS:
Drug: Apixaban 2.5 MG Oral Tablet [ELIQUIS] — Apixaban 5 MG BID versus Apixaban 2.5 MG BID
  Other Names: Apixaban 5 MG Oral Tablet

SUMMARY:
Isolated distal DVT (iDDVT) is the most frequent clinical presentation of VTE and is associated with a significant morbidity and risks of long-term complications. Data from clinical trials highlighted that patients with iDDVT might require some level of AC treatment. However, the optimal anticoagulant intensity is uncertain, and it is plausible that the best benefit/risk ratio for AC might be achieved with lower intensity doses rather than therapeutic doses.

The principal research question of the Apixaban to treat calf vein thrombosis (API-CALF) study is to determine whether, after a conventional course of 7 days of Apixaban 10mg BID, Apixaban 2.5mg BID (experimental arm) is non inferior to Apixaban 5 mg BID (standard arm) in preventing VTE recurrence and bleeding in patients with iDDVT. Patients will be treated with Apixaban for a total of 3 months. In that perspective we will conduct an international multicentre open-label assessor-blinded study

DETAILED DESCRIPTION:
Isolated distal deep vein thrombosis (iDDVT) is an infra-popliteal DVT, without concomitant proximal DVT and without pulmonary embolism (PE). Until recently, few large studies have focused on iDDVT, and the clinical significance and therapeutic management of iDDVT was mostly based on expert opinion and "gestalt" rather than on strong scientific data. iDDVT is the most frequent presentation of venous thromboembolic disease (VTE). Indeed, in the large French, multicentre, observational, OPTIMEV study, where all patients with suspected DVT underwent systematic whole leg compression ultrasound (CUS) exploration, iDDVT represented 56% of all DVTs. A similar high proportion of distal DVT among DVT (52.1%) was reported in Johnson's meta-analysis.

The risk of proximal extension of iDDVT to the proximal veins is substantial. In an extensive review of the literature published 15 years ago, the investigators reported that the risk of proximal extension of iDDVT, whether treated or left untreated, ranged from 0-44%, underlining the heterogeneity of the available data. Data from the CALTHRO study and CACTUS trial and extrapolation of data from management studies comparing the safety of serial proximal CUS vs. whole leg CUS for DVT diagnosis suggest that the rate of extension of untreated iDDVT to proximal deep veins was ~ 10% and up to 28% in high-risk populations, such as patients with cancer (3, 7-9). This 10% average risk of proximal extension is far above the usual 2% cut-off for an acceptable false-negative rate for negative findings in DVT diagnostic strategies. Hence, from a strict natural history standpoint, clinical significance of iDDVT is no longer in question. In summary, iDDVT is the most frequent clinical presentation of VTE and patients with iDDVT are at significant risk of proximal extension and of adverse outcomes both in the short and in the long-term.

Management of iDDVT is one of the most debated issue in the field of VTE. Thus, in all trials that validated the use of DOAC, distal location of DVT was an exclusion criterion.

While the American society of Hematology (ASH) guidelines do not comment on iDDVT specific treatment, the American college of chest physicians (ACCP) guidelines state that only 'high risk' distal DVT should be systematically treated with anticoagulation. Non high risk iDDVT could benefit from surveillance by repeated CUS. However, in the international CACTUS study, the investigators observed that a primary reason for refusal of participation and failure to fulfil recruitment was that patients and their treating physicians refused that iDDVT be left untreated. In routine clinical practice, data from observational registries showed that the majority iDDVT are treated with full dose of anticoagulants: 97% of iDDVT in the French OPTIMEV study, 98% in the Italian MASTER registry and 99% in the international RIETE registry. These therapeutic attitudes reflect physicians' beliefs (and patients' preference) that anticoagulation is important in case of iDDVT.

For proximal DVT and PE, "therapeutic" doses of anticoagulants are prescribed as use of lower doses was associated with an unacceptably high VTE risk. In contrast, for superficial vein thrombosis (SVT), "prophylactic" doses (fondaparinux 2.5mg or rivaroxaban 10 mg daily) were shown to be very effective and associated with a very low bleeding risk. Regarding iDDVT, risk of VTE recurrence and effectiveness of different dose regimen of anticoagulation are less clear and literature suggests that it could depend on patients' characteristics . Based on literature review, main risk factors for VTE extension/recurrence include cancer, calf trifurcation involvement, previous VTE, unprovoked character of DVT or presence of a permanent risk factor, and multiple vein distal vein thromboses.

In the CACTUS study, at 3 months, the proportion of extension to proximal deep veins in the therapeutic anticoagulation arm was lower than in the placebo arm (3.3% vs. 6.2% at 3 months; p=NS), but the risk of significant bleeding was significantly higher (4.1% vs. 0.0%)(3). Namely, in CACTUS, the benefit of therapeutic anticoagulation in terms of VTE risk reduction was offset by the excess in risk of bleeding.

In summary, iDDVT is the most frequent clinical presentation of VTE and is associated with a significant morbidity and risks of long-term complications. Data from clinical trials highlighted that patients with iDDVT might require some level of AC treatment. However, the optimal anticoagulant intensity is uncertain, and it is plausible that the best benefit/risk ratio for AC might be achieved with lower intensity doses rather than therapeutic doses.

The principal research question of the Apixaban to treat calf vein thrombosis (API-CALF) study is to determine whether, after a conventional course of 7 days of Apixaban 10mg BID, Apixaban 2.5mg BID (experimental arm) is non inferior to Apixaban 5 mg BID (standard arm) in preventing VTE recurrence and bleeding in patients with iDDVT. Patients will be treated with Apixaban for a total of 3 months. In that perspective we will conduct an international multicentre open-label assessor-blinded study

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients with acute (symptoms <10 days) symptomatic iDDVT diagnosed on leg CUS who have none of the following exclusion criteria and who provided informed consent to participate. Diagnosis of iDDVT is made in the presence of an incompressible distal deep vein (deep calf vein (posterior tibial, anterior tibial or peroneal veins) or muscular vein (soleal or gastrocnemius veins)).

Exclusion Criteria:

* Age < 18 years
* Ipsi or contralateral Proximal DVT
* Distal DVT involving the tibio-peroneal trunk (i.e. calf trifurcation)
* DVT occurring while on anticoagulation (started ≥48hours before DVT diagnosis); However, inpatients that developed their iDDVT while on prophylactic anticoagulation are eligible if their expected date of discharge is <6 days post randomization.
* Clinically suspected PE (patient eligible if PE ruled out with objective tests)
* Active cancer, receiving cancer treatment or cured for < 6 months
* Indication for long-term therapeutic anticoagulation (e.g. atrial fibrillation, mechanical heart valve…)
* Thrombocytopenia (platelet count <100 g/l)
* Severe renal impairment (creatinine clearance <30 ml/min)
* Liver disease (including Child-Pugh Class B and C) associated with coagulopathy
* Pregnant or breast-feeding woman
* Body weight >120kg or <40 kg
* Ongoing active bleeding or condition at high risk of bleeding with anticoagulation (e.g. peptic ulcer…)
* Treatment with daily NSAIDs (aspirin ≤160 mg/day or clopidogrel ≤75 mg day permitted)
* Allergy to Apixaban
* Use of concomitant drugs that significantly interact with Apixaban: strong inhibitors of P-gp and CYP3A4 or strong inducers of CYP3A4
* Treatment with anticoagulants at therapeutic dose >2 days after DVT diagnosis
* Life expectancy < 1 year
* Enrolled in another clinical trial within previous 30 days
* Inability or refusal to provide informed consent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of i) symptomatic VTE; ii) major bleeding and clinically relevant non major bleeding (CRNMB); iii) VTE and bleeding related death. | 1 year
  The primary outcome is a composite of rate of i) symptomatic VTE (includes iDDVT involving a new distal deep vein, proximal DVT or PE; ii) major bleeding and clinically relevant non major bleeding (CRNMB); iii) VTE and bleeding related death.

SECONDARY OUTCOMES:
Individual components of the composite endpoint at 3 months and 1 year - Generic and venous disease-specific QOL scores at 1 year - Patient's compliance with treatment at 3 months - Serious adverse events during follow-up - PTS as measured at 1 year | 1 year
  as above
Generic and venous disease-specific QOL scores at 1 year | 1 year
  QOL score
Patient's observance with treatment at 3 months | 3 months
  Observance of the patient
Serious adverse events during follow-up | 1 year
  Adverse events
PTS as measured at 1 year | 1 year
  Post thrombotic syndrome assessed with the Villalta scale

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Galanaud, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre and University of Toronto, Toronto, Canada; Marc Righini, MD, Principal Investigator — Geneva University Hospital, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual research subjects' data cannot legally nor ethically be made available to non authorised people (HRA, cf. §7). According to the research subjects' informed consent, only the sponsor, the investigation team, reviewers, auditors and inspection authorities are entitled to access such data.

REFERENCES:
- [Result] Galanaud JP, Bosson JL, Quere I. Risk factors and early outcomes of patients with symptomatic distal vs. proximal deep-vein thrombosis. Curr Opin Pulm Med. 2011 Sep;17(5):387-91. doi: 10.1097/MCP.0b013e328349a9e3. PMID 21832920
- [Result] Schellong SM. Distal DVT: worth diagnosing? Yes. J Thromb Haemost. 2007 Jul;5 Suppl 1:51-4. doi: 10.1111/j.1538-7836.2007.02490.x. PMID 17635708
- [Result] Righini M, Galanaud JP, Guenneguez H, Brisot D, Diard A, Faisse P, Barrellier MT, Hamel-Desnos C, Jurus C, Pichot O, Martin M, Mazzolai L, Choquenet C, Accassat S, Robert-Ebadi H, Carrier M, Le Gal G, Mermilllod B, Laroche JP, Bounameaux H, Perrier A, Kahn SR, Quere I. Anticoagulant therapy for symptomatic calf deep vein thrombosis (CACTUS): a randomised, double-blind, placebo-controlled trial. Lancet Haematol. 2016 Dec;3(12):e556-e562. doi: 10.1016/S2352-3026(16)30131-4. Epub 2016 Nov 8. PMID 27836513
- [Result] Galanaud JP, Sevestre-Pietri MA, Bosson JL, Laroche JP, Righini M, Brisot D, Boge G, van Kien AK, Gattolliat O, Bettarel-Binon C, Gris JC, Genty C, Quere I; OPTIMEV-SFMV Investigators. Comparative study on risk factors and early outcome of symptomatic distal versus proximal deep vein thrombosis: results from the OPTIMEV study. Thromb Haemost. 2009 Sep;102(3):493-500. doi: 10.1160/TH09-01-0053. PMID 19718469
- [Result] Johnson SA, Stevens SM, Woller SC, Lake E, Donadini M, Cheng J, Labarere J, Douketis JD. Risk of deep vein thrombosis following a single negative whole-leg compression ultrasound: a systematic review and meta-analysis. JAMA. 2010 Feb 3;303(5):438-45. doi: 10.1001/jama.2010.43. PMID 20124539
- [Result] Righini M, Bounameaux H. Clinical relevance of distal deep vein thrombosis. Curr Opin Pulm Med. 2008 Sep;14(5):408-13. doi: 10.1097/MCP.0b013e32830460ea. PMID 18664970
- [Result] Palareti G, Cosmi B, Lessiani G, Rodorigo G, Guazzaloca G, Brusi C, Valdre L, Conti E, Sartori M, Legnani C. Evolution of untreated calf deep-vein thrombosis in high risk symptomatic outpatients: the blind, prospective CALTHRO study. Thromb Haemost. 2010 Nov;104(5):1063-70. doi: 10.1160/TH10-06-0351. Epub 2010 Aug 5. PMID 20694281
- [Result] Bernardi E, Camporese G, Buller HR, Siragusa S, Imberti D, Berchio A, Ghirarduzzi A, Verlato F, Anastasio R, Prati C, Piccioli A, Pesavento R, Bova C, Maltempi P, Zanatta N, Cogo A, Cappelli R, Bucherini E, Cuppini S, Noventa F, Prandoni P; Erasmus Study Group. Serial 2-point ultrasonography plus D-dimer vs whole-leg color-coded Doppler ultrasonography for diagnosing suspected symptomatic deep vein thrombosis: a randomized controlled trial. JAMA. 2008 Oct 8;300(14):1653-9. doi: 10.1001/jama.300.14.1653. PMID 18840838
- [Result] Gibson NS, Schellong SM, Kheir DY, Beyer-Westendorf J, Gallus AS, McRae S, Schutgens RE, Piovella F, Gerdes VE, Buller HR. Safety and sensitivity of two ultrasound strategies in patients with clinically suspected deep venous thrombosis: a prospective management study. J Thromb Haemost. 2009 Dec;7(12):2035-41. doi: 10.1111/j.1538-7836.2009.03635.x. Epub 2009 Oct 8. PMID 19817986
- [Result] Bates SM, Jaeschke R, Stevens SM, Goodacre S, Wells PS, Stevenson MD, Kearon C, Schunemann HJ, Crowther M, Pauker SG, Makdissi R, Guyatt GH. Diagnosis of DVT: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e351S-e418S. doi: 10.1378/chest.11-2299. PMID 22315267
- [Result] Galanaud JP, Sevestre MA, Genty C, Pernod G, Quere I, Bosson JL. Is it useful to also image the asymptomatic leg in patients with suspected deep vein thrombosis?: comment. J Thromb Haemost. 2015 Nov;13(11):2127-30. doi: 10.1111/jth.13123. Epub 2015 Sep 30. No abstract available. PMID 26332772
- [Result] Palareti G. How I treat isolated distal deep vein thrombosis (IDDVT). Blood. 2014 Mar 20;123(12):1802-9. doi: 10.1182/blood-2013-10-512616. Epub 2014 Jan 28. PMID 24472834
- [Result] Palareti G, Schellong S. Isolated distal deep vein thrombosis: what we know and what we are doing. J Thromb Haemost. 2012 Jan;10(1):11-9. doi: 10.1111/j.1538-7836.2011.04564.x. PMID 22082302
- [Result] Righini M. Is it worth diagnosing and treating distal deep vein thrombosis? No. J Thromb Haemost. 2007 Jul;5 Suppl 1:55-9. doi: 10.1111/j.1538-7836.2007.02468.x. PMID 17635709
- [Result] Masuda EM, Kistner RL, Musikasinthorn C, Liquido F, Geling O, He Q. The controversy of managing calf vein thrombosis. J Vasc Surg. 2012 Feb;55(2):550-61. doi: 10.1016/j.jvs.2011.05.092. Epub 2011 Oct 26. PMID 22032881
- [Result] Lohr JM, Fellner AN. Isolated calf vein thrombosis should be treated with anticoagulation. Dis Mon. 2010 Oct;56(10):590-600. doi: 10.1016/j.disamonth.2010.06.010. No abstract available. PMID 20971330
- [Result] Masuda EM, Kistner RL. The case for managing calf vein thrombi with duplex surveillance and selective anticoagulation. Dis Mon. 2010 Oct;56(10):601-13. doi: 10.1016/j.disamonth.2010.06.011. No abstract available. PMID 20971331
- [Result] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Masiukiewicz U, Pak R, Thompson J, Raskob GE, Weitz JI; AMPLIFY Investigators. Oral apixaban for the treatment of acute venous thromboembolism. N Engl J Med. 2013 Aug 29;369(9):799-808. doi: 10.1056/NEJMoa1302507. Epub 2013 Jul 1. PMID 23808982
- [Result] Bauersachs RM, Herold J. Oral Anticoagulation in the Elderly and Frail. Hamostaseologie. 2020 Feb;40(1):74-83. doi: 10.1055/s-0040-1701476. Epub 2020 Jan 30. PMID 32000266
- [Result] Schulman S, Kearon C, Kakkar AK, Schellong S, Eriksson H, Baanstra D, Kvamme AM, Friedman J, Mismetti P, Goldhaber SZ; RE-MEDY Trial Investigators; RE-SONATE Trial Investigators. Extended use of dabigatran, warfarin, or placebo in venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):709-18. doi: 10.1056/NEJMoa1113697. PMID 23425163
- [Result] Hokusai-VTE Investigators; Buller HR, Decousus H, Grosso MA, Mercuri M, Middeldorp S, Prins MH, Raskob GE, Schellong SM, Schwocho L, Segers A, Shi M, Verhamme P, Wells P. Edoxaban versus warfarin for the treatment of symptomatic venous thromboembolism. N Engl J Med. 2013 Oct 10;369(15):1406-15. doi: 10.1056/NEJMoa1306638. Epub 2013 Aug 31. PMID 23991658
- [Result] EINSTEIN-PE Investigators; Buller HR, Prins MH, Lensin AW, Decousus H, Jacobson BF, Minar E, Chlumsky J, Verhamme P, Wells P, Agnelli G, Cohen A, Berkowitz SD, Bounameaux H, Davidson BL, Misselwitz F, Gallus AS, Raskob GE, Schellong S, Segers A. Oral rivaroxaban for the treatment of symptomatic pulmonary embolism. N Engl J Med. 2012 Apr 5;366(14):1287-97. doi: 10.1056/NEJMoa1113572. Epub 2012 Mar 26. PMID 22449293
- [Result] Kearon C, Akl EA, Ornelas J, Blaivas A, Jimenez D, Bounameaux H, Huisman M, King CS, Morris TA, Sood N, Stevens SM, Vintch JRE, Wells P, Woller SC, Moores L. Antithrombotic Therapy for VTE Disease: CHEST Guideline and Expert Panel Report. Chest. 2016 Feb;149(2):315-352. doi: 10.1016/j.chest.2015.11.026. Epub 2016 Jan 7. PMID 26867832
- [Result] Ortel TL, Neumann I, Ageno W, Beyth R, Clark NP, Cuker A, Hutten BA, Jaff MR, Manja V, Schulman S, Thurston C, Vedantham S, Verhamme P, Witt DM, D Florez I, Izcovich A, Nieuwlaat R, Ross S, J Schunemann H, Wiercioch W, Zhang Y, Zhang Y. American Society of Hematology 2020 guidelines for management of venous thromboembolism: treatment of deep vein thrombosis and pulmonary embolism. Blood Adv. 2020 Oct 13;4(19):4693-4738. doi: 10.1182/bloodadvances.2020001830. PMID 33007077
- [Result] Palareti G, Agnelli G, Imberti D, Moia M, Ageno W, Pistelli R, Rossi R, Verso M; MASTER Investigators. Do Italian vascular centers look for isolated calf deep vein thrombosis? Analysis of isolated calf deep vein thromboses included in the ''Master'' Registry. Int Angiol. 2008 Dec;27(6):482-8. PMID 19078910
- [Result] Galanaud JP, Trujillo-Santos J, Bikdeli B, Di Micco P, Bortoluzzi C, Bertoletti L, Pedrajas JM, Ballaz A, Alfonso J, Monreal M; RIETE Investigators. Management of isolated distal deep-vein thrombosis with direct oral anticoagulants in the RIETE registry. J Thromb Thrombolysis. 2021 Aug;52(2):532-541. doi: 10.1007/s11239-020-02347-6. Epub 2020 Nov 28. PMID 33247808
- [Result] Hull R, Delmore T, Genton E, Hirsh J, Gent M, Sackett D, McLoughlin D, Armstrong P. Warfarin sodium versus low-dose heparin in the long-term treatment of venous thrombosis. N Engl J Med. 1979 Oct 18;301(16):855-8. doi: 10.1056/NEJM197910183011602. PMID 384248
- [Result] Decousus H, Prandoni P, Mismetti P, Bauersachs RM, Boda Z, Brenner B, Laporte S, Matyas L, Middeldorp S, Sokurenko G, Leizorovicz A; CALISTO Study Group. Fondaparinux for the treatment of superficial-vein thrombosis in the legs. N Engl J Med. 2010 Sep 23;363(13):1222-32. doi: 10.1056/NEJMoa0912072. PMID 20860504
- [Result] Beyer-Westendorf J, Schellong SM, Gerlach H, Rabe E, Weitz JI, Jersemann K, Sahin K, Bauersachs R; SURPRISE investigators. Prevention of thromboembolic complications in patients with superficial-vein thrombosis given rivaroxaban or fondaparinux: the open-label, randomised, non-inferiority SURPRISE phase 3b trial. Lancet Haematol. 2017 Mar;4(3):e105-e113. doi: 10.1016/S2352-3026(17)30014-5. Epub 2017 Feb 16. PMID 28219692
- [Result] Quere I, Elias A, Maufus M, Elias M, Sevestre MA, Galanaud JP, Bosson JL, Bura-Riviere A, Jurus C, Lacroix P, Zuily S, Diard A, Wahl D, Bertoletti L, Brisot D, Frappe P, Gillet JL, Ouvry P, Pernod G. [Unresolved questions on venous thromboembolic disease. Consensus statement of the French Society for Vascular Medicine (SFMV)]. J Med Vasc. 2019 Feb;44(1):e1-e47. doi: 10.1016/j.jdmv.2018.12.178. Epub 2019 Feb 2. No abstract available. French. PMID 30770089
- [Result] Galanaud JP, Sevestre MA, Pernod G, Kahn SR, Genty C, Terrisse H, Brisot D, Gillet JL, Quere I, Bosson JL. Long-term risk of venous thromboembolism recurrence after isolated superficial vein thrombosis. J Thromb Haemost. 2017 Jun;15(6):1123-1131. doi: 10.1111/jth.13679. Epub 2017 May 5. PMID 28317330